CLINICAL TRIAL: NCT03164525
Title: Validation of the Thai Version Critical Care Pain Observation Tool and Behavioral Pain Scale in Postoperative Mechanically Ventilated ICU Patients
Brief Title: Validation of the Thai Version CPOT and BPS in Postoperative ICU Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Karuna Wongtangman, MD, Mahidol University
Other Study IDs: Si553/2014
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Adult ICU Patients
Keywords: Thai version; validated; Critical Care Pain Observation Tool; Behavioral Pain Scale; adult ICU patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Critical care pain observation tool (CPOT) — test validity and reliability of Thai-version CPOT and BPS
  Other Names: Behavioral pain scale (BPS)

SUMMARY:
The prospective study set forth to test Thai version CPOT and BPS for validity, reliability, and practicality. After translation, both pain scales were tested for concurrent validity, discriminant validity, criterion validity, and inter-rater reliability in patients who were intubated during the postoperative period. Opinions regarding practicality were elicited via questionnaires from nurses who had been using and were familiar with these two pain scales.

DETAILED DESCRIPTION:
The prospective study set forth to test Thai version CPOT and BPS for validity, reliability, and practicality. After translation, both pain scales were tested for concurrent validity, discriminant validity, criterion validity, and inter-rater reliability in patients who were intubated during the postoperative period. Opinions regarding practicality were elicited via questionnaires from nurses who had been using and were familiar with these two pain scales.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years
* be able to communicate in Thai
* intubated during postoperative period.

Exclusion Criteria:

* quadriplegia
* patients with limb or facial injuries
* patients receiving neuromuscular blockers
* patients with limb mobility adversely affected by stroke
* patients with epidural catheter used for postoperative pain control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative Mechanically Ventilated Adult ICU Patients
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
construct validity | before and after analgesic given during 24 hours postoperative period

SECONDARY OUTCOMES:
content validity, concurrent validity, inter-rater reliability, and practicality | 24 hours after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No